CLINICAL TRIAL: NCT02728531
Title: A Pilot Study of Bendamustine and Rituximab Alternating With Cytarabine and Rituximab for Untreated Mantle Cell Lymphoma
Brief Title: Bendamustine and Rituximab Alternating With Cytarabine and Rituximab for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201603149
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab; Cytarabine; pegfilgrastim; Granulocyte Colony-Stimulating Factor; Leukapheresis; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bendamustine, Rituximab, Cytarabine (Experimental): * Bendamustine on Days 1 and 2 of Cycles 1, 3, and 5.
  * In Cycle 1, rituximab on Day 1 or 2 at the investigator's discretion. Given on Day 1 of Cycles 2 through 6.
  * On Days 1 and 2 of Cycles 2, 4, and 6, cytarabine will be administered every 12 hours for a total of 4 doses.
  * Growth factor will be administered subcutaneously within 72 hours of completion of each even-numbered cycles of chemotherapy.
  * Leukapheresis will begin when the total WBC ≥ 5000/ μL and continue daily until collection of ≥ 2x106 CD34+ cells/kg (with a maximum of 5 courses of apheresis).
  * Standard of care peripheral blood autologous stem cell harvest will proceed per institutional guidelines and begin during Cycle 6 following rituximab and cytarabine therapy, when the total WBC ≥ 5000/ μL. Collection will continue on a daily basis until collection of ≥ 2x106 CD34+ cells/kg.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Cytarabine; Drug: Pegfilgrastim; Procedure: Leukapheresis; Drug: Filgrastim; Procedure: Autologous stem cell transplant

INTERVENTIONS:
Drug: Bendamustine
  Other Names: Bendamustine Hydrochloride; Treanda
Drug: Rituximab
  Other Names: Rituxan
Drug: Cytarabine
  Other Names: Cytosar-U; Tarabine PFS
Drug: Pegfilgrastim
  Other Names: Neulasta; G-CSF
Procedure: Leukapheresis
Drug: Filgrastim
  Other Names: Neupogen
Procedure: Autologous stem cell transplant

SUMMARY:
Given the established role of high dose cytarabine (HiDAC) combined with rituximab, along with recent data showing the encouraging efficacy of bendamustine, the investigators seek to integrate the synergistic effects of these medicines in alternating cycles as induction therapy prior to autologous stem cell transplant (ASCT). Based on prior experience with bendamustine and rituximab (BR) based induction therapy, the investigators seek to evaluate the efficacy and safety of stem cell mobilization in this pilot study

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell lymphoma with documented expression of CD20 (or CD 19) and cyclin D1 (BCL1) by immunohistochemical stains and/or t (11; 14) by cytogenetics or FISH
* Eighteen to 65 years of age, inclusive.
* Presence of evaluable disease by PET imaging per the Lugano classification (Cheson 201418)
* Eligible for autologous stem cell transplantation.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcl unless in the opinion of the treating physician, neutropenia is due to splenomegaly or bone marrow involvement
  * Platelets ≥ 100,000/mcl unless in the opinion of the treating physician, thrombocytopenia is due to splenomegaly or bone marrow involvement
  * Total bilirubin ≤ 2 x IULN and AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN except when, in the opinion of the treating physician, is due to direct involvement of lymphoma (e.g., hepatic infiltration or biliary obstruction due to lymphoma) or Gilbert's disease
  * Creatinine ≤ IULN OR creatinine clearance ≥ 40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Negative HIV serology.

Exclusion Criteria:

* Any previous chemotherapy or radiation for mantle cell lymphoma. Short course of steroids for symptom relief prior to presentation is permissible.
* Symptomatic meningeal or parenchymal brain lymphoma.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab, cytarabine, bendamustine or other agents used in the study.
* Severe concurrent illness, which would limit compliance with study requirements.
* Subjects with serologic status reflecting active viral hepatitis B or C infection are not eligible. Subjects whoare hepatitis B core antibody positive but antigen negative will need negative polymerase chain reaction (PCR) prior to enrollment. Hepatitis B surface antigen positive or PCR positive patients will be excluded. Subjects who are hepatitis C antibody positive will need negative PCR prior to enrollment. Patients with positive hepatitis C will be excluded.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Stem cell mobilization success rate | Completion of stem cell mobilization (approximately 25 weeks)
  -Stem cell mobilization success is defined as a yield of ≥ 2 x 106 CD34+ stem cells/kg with a maximum of 5 courses of apheresis.

SECONDARY OUTCOMES:
Overall response rate | Completion of treatment (approximately 24 weeks)
  -Response to treatment is guided based upon the Recommendations for Initial Evaluation, Staging and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.
Pre-transplant complete response rate (CRR) | Completion of treatment (approximately 24 weeks)
  CRR=
  * Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  * London Deauville score of 1 and 2 in lymph nodes and extra lymphatic sites is considered to represent complete metabolic response. A London Deauville score 3 in the post treatment PET scan may be considered to represent complete metabolic response especially if it is not higher than the surrounding normal physiologic uptake.
  * No evidence of FDG avid disease in the bone marrow
  * No new lesions
  * If the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
Progression-free survival (PFS) | 5 years
  -PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | 5 years
Safety and tolerability of bendamustine and rituximab alternating with cytarabine and rituximab as measured by grades 3 or higher toxicities | 30 days following completion of treatment (approximately 29 weeks)
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merryman RW, Edwin N, Redd R, Bsat J, Chase M, LaCasce A, Freedman A, Jacobson C, Fisher D, Ng S, Crombie J, Kim A, Odejide O, Davids MS, Brown JR, Jacene H, Cashen A, Bartlett NL, Mehta-Shah N, Ghobadi A, Kahl B, Joyce R, Armand P, Jacobsen E. Rituximab/bendamustine and rituximab/cytarabine induction therapy for transplant-eligible mantle cell lymphoma. Blood Adv. 2020 Mar 10;4(5):858-867. doi: 10.1182/bloodadvances.2019001355. PMID 32126141
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu